CLINICAL TRIAL: NCT06670352
Title: A Randomized, Double-blind, and Placebo-controlled Parallel Phase II Clinical Study to Evaluate the Efficacy and Safety of HSK39297 Tablets in Treatment of Patients with Primary IgAN
Brief Title: Phase II Study of Efficacy and Safety of HSK39297 Tablet in Treatment of Patients with Primary IgAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK39297-202
Record Dates: First submitted 2024-10-15; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: IgA Nephropathy (IgAN)
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- HSK39297 50mg BID (Experimental)
  Interventions: Drug: HSK39297 50mgBID
- HSK39297 100mg BID (Experimental)
  Interventions: Drug: HSK39297 100mgBID
- HSK39297 200mg QD (Experimental)
  Interventions: Drug: HSK39297 200mgQD

INTERVENTIONS:
Drug: Placebo — QD or BID, 24-weeks fixed dose.
  Arms: Placebo
Drug: HSK39297 50mgBID — 24-weeks fixed dose.
  Arms: HSK39297 50mg BID
Drug: HSK39297 100mgBID — 24-weeks fixed dose.
  Arms: HSK39297 100mg BID
Drug: HSK39297 200mgQD — 24-weeks fixed dose.
  Arms: HSK39297 200mg QD

SUMMARY:
Evaluate the efficacy and safety of HSK39297 tablets in patients with primary IgAN

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed and dated an IRB/IEC approved written informed consent form.Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study.
2. Female and male patients above 18 years of age.
3. Patients must weigh at least 35 kg to participate in the study, and must have a body mass index (BMI) below 35 kg/m2. BMI = Body weight (kg) / [Height (m)]2
4. Subjects with a biopsy-verified IgA nephropathy and where the biopsy was performed within the prior five years.
5. Urine protein ≥0.75g/24hr or FMV UPCR≥0.8g/g at screening.
6. Measured Glomerular Filtration Rate (GFR) or estimated GFR (using the CKD-EPI formula 2021) ≥30 mL/min per 1.73 m2.

Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 90 days, whichever is longer.
2. All transplanted patients (any organ, including bone marrow).
3. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
4. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study.
5. Pregnant or nursing (lactating) women.
6. Plasma donation (≥ 400mL) within 12 weeks prior to first dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-11-23 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
The ratio of 24-hour urine protein to creatinine (24h-UPCR) compared to baseline after 12 weeks of treatment | From week 1 to week 12

SECONDARY OUTCOMES:
The ratio of 24-hour urine protein to creatinine (24h-UPCR) compared to baseline after 24 weeks of treatment | From week 1 to week 24
The ratio of 24h-UPCR compared to baseline at each clinical visit point during the treatment period | From week 1 to week 24
The ratio of 24-hour urine protein (24h-UPE) compared to baseline at each clinical visit point during the treatment period | From week 1 to week 24
The change in estimated glomerular filtration rate (eGFR, CKD-EPI 2021 formula) compared to baseline at each clinical visit point during the treatment period | From week 1 to week 24
The change in blood creatinine compared to baseline at each clinical visit point during the treatment period | From week 1 to week 24
The ratio of FMV UPCR, urinary albumin to creatinine ratio (UACR) compared to baseline at each clinical visit point during the treatment period | From week 1 to week 24
The change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale score compared to baseline at each clinical visit point during the treatment period | From week 1 to week 24
  0-52, the higher the score, the better the QOL.
Incidence , severity and relationship of adverse events during the study period | From week 1 to week 24
Plasma Pharmacokinetics (PK) of Time to Maximum Concentration at Steady State (Tmax,ss) of HSK39297 | From week 1 to week 24
Plasma Pharmacokinetics (PK) of Area Under the Curve at Steady State (AUCtau,ss and AUClast,ss) of HSK39297 | From week 1 to week 24
Plasma Pharmacokinetics (PK) of Pre-dose Trough at Steady State (Ctrough,ss) of HSK39297 | From week 1 to week 24
Plasma Pharmacokinetics (PK) of Maximum Concentrations (Cmax,ss) at Steady State of HSK39297 | From week 1 to week 24
Changes in alternative pathway (AP) complement activity compared to baseline at each clinical visit point during the treatment period | From week 1 to week 24
Changes in plasma Bb levels compared to baseline at each clinical visit point during the treatment period | From week 1 to week 24
Changes in plasma and urine sC5b-9 levels compared to baseline at each clinical visit point during the treatment period | From week 1 to week 24

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu